CLINICAL TRIAL: NCT02458599
Title: A Study to Evaluate the Effects of Protein Supplementation in Attenuating the Decline in Performance Following Strenuous Concurrent Exercise
Brief Title: Efficacy Study of Protein Supplementation in Attenuating the Decline in Performance After Strenuous Concurrent Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 204676
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Sports Nutritional Sciences

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test product (Experimental): One ready-to-drink beverage of 500 milliliter (mL) volume, containing 20 gram (g) protein will be administered orally, twice daily for four days.
  Interventions: Dietary Supplement: Test product
- Reference product 1 (Active Comparator): One ready-to-drink beverage of 500 mL volume, containing 20 g carbohydrate will be administered orally, twice daily for four days.
  Interventions: Dietary Supplement: Reference product 1
- Reference product 2 (Placebo Comparator): One ready-to-drink beverage of 500 mL volume, containing 0 g carbohydrate will be administered orally, twice daily for four days.
  Interventions: Dietary Supplement: Reference product 2

INTERVENTIONS:
Dietary Supplement: Test product — Whey protein hydrolysate (20 g)
  Arms: Test product
Dietary Supplement: Reference product 1 — Iso-energetic carbohydrate (20 g)
  Arms: Reference product 1
Dietary Supplement: Reference product 2 — Negligible energy placebo (20 g)
  Arms: Reference product 2

SUMMARY:
This study is designed to investigate whether protein supplementation can improve recovery of muscle function following a strenuous combination of both endurance and resistance exercise. It will specifically investigate the effect of protein supplementation on the recovery of strength, power and endurance exercise performance, along with measures of damage and inflammation of the muscle.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary informed consent form and has received signed and dated copy of the informed consent form
* Male participants; age between 18 to 35 years, inclusive
* Well trained endurance cyclist (competing at a minimum of Category 3 road-racing/estimated 10 mile TT of <23 minutes), with a training history >1 year
* Good general and mental health

Exclusion Criteria:

* Currently taking any nutritional supplements, polyphenols or beta-blockers, Non-steroidal anti-inflammatory drugs (NSAIDs), recreational drugs
* Known or suspected intolerance or hypersensitivity to the study material or any of their stated ingredients
* Allergy to milk or wheat products
* Heart or any other medical condition that may contra-indicate participants from taking part in high intensity or exhaustive physical activity
* Previous participation in this study; another clinical study or receipt of an investigational drug within 30 days of the screening visit; participation in another study involving a protocol to elicit Exercise-Induced Muscle Damage (EIMD) within 6 months of the screening visit

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Isometric Maximal Voluntary Contraction (MVC) Assessment | 96 hours (h)
  Maximum voluntary isometric contraction (MVIC) will be assessed at the knee during a leg extension movement using an isokinetic dynamometer. MVIC will be used to assess strength. Participants will perform the exercise using the dominant leg at a knee joint angle of 70º three times, with a contraction of 3 seconds (s) on each occasion (each contraction separated by 60 s rest). The peak force (measured in Newton) generated across the three repetitions will be recorded.
Counter Movement Jump (CMJ) Assessment | 96 h
  Power will be assessed using counter-movement jump. Participants will place their hands on their hips, descend rapidly to ~90º knee joint angle, and then jump as high as possible using a counter-movement. Three jumps will be performed (each jump separated by 60 s rest) and the peak vertical jump height (measured in centimeters) will be recorded.
16.1 Kilometer (km) Cycling Time Trial (TT) Assessment | 96 h
  The 16.1 km cycling TT assessment will be performed on a cycling ergometer. Participants will be required to complete a distance of 16.1 km in as short a time as possible, while being blinded to time elapsed.

SECONDARY OUTCOMES:
Serum Creatine Kinase Analysis | 96 h
  Muscle damage will be assessed by analyzing serum creatine kinase (CK) using CK N-Acetyl-L Cysteine (NAC)-activated Enzyme Linked Immunosorbent Assay (ELISA).
Serum C-Reactive Protein Analysis | 96 h
  Muscle inflammation will be assessed by analyzing serum high sensitivity (hs) C-reactive protein (CRP) using hs-CRP ELISA.
Perceived Muscle Soreness Assessment | 96 h
  Perceived muscle soreness will be measured on a 200 mm visual analogue scale (VAS) where 0 mm= no pain and 200 mm= unbearably painful. Participants will be required to hold a fixed squat position (90º knee joint angle) while perceived muscle soreness is rated.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Brentford, United Kingdom